CLINICAL TRIAL: NCT02975804
Title: Effectiveness of Interactive Computer Play on Trunk Control and Gross Motor Function in Children With Cerebral Palsy: a Pilot Randomized Controlled Trial
Brief Title: RCT on Interactive Computer Play on Trunk Control in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Tamis Wai-mun PIN, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14150171
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Cerebral Palsy; Exercise Therapy; Postural Balance
Keywords: cerebral palsy; video games; postural control; balance; children
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive computer play (ICP) (Experimental): The children in the treatment group will receive training on their trunk control using the Tymo in sitting 4 times per week for 20 minutes per session. The treatment will last for 6 weeks. All study children will continue their usual therapies at school.
  Interventions: Device: Tymo
- Standard Therapy (No Intervention): Children in the control group will continue their usual therapy.

INTERVENTIONS:
Device: Tymo — All children will be calibrated using the Tymo in a static sitting position in each treatment session. The amplitude of the force and weight distribution generated by the child between the two sides of the body will be recorded. This information will be used to set up the Tymo as a training module (the intervention) by the software, in which the child will move the trunk forward, backward and sideways to participate in a computer game in sitting. The child will choose which game they want in each treatment session and they have to stay on the same game for at least 10 minutes before changing to another game.
  Arms: Interactive computer play (ICP)

SUMMARY:
Objectives:

This proposal is to investigate the effect of a 6-week training programme using an Interactive computer play (ICP) on the trunk control, balance and gross motor function in children with cerebral palsy (CP).

Hypothesis to be tested:

The trunk control, balance and gross motor function of children with CP will be significantly improved after the ICP programme.

Design and subjects:

20 children (6 to 12 years old) with CP will be recruited in this pilot randomised controlled trial. The children will be randomly allocated into a control or treatment group (10 children in each arm).

Study instruments:

Tymo is a wireless force plate used for assessment and training.

Intervention:

An ICP program will be set up using the Tymo. The child uses their trunk movements in the ICP in sitting during the intervention. The children will receive the intervention 4 times/week, 20 minutes/session for 6 weeks. All children will be assessed at the beginning, 3, 6 and 12 weeks post-intervention.

Main outcome measures:

* Segmental Assessment on Trunk control
* Pediatric Reach Test
* Gross Motor Function Measure Item Set (GMFM IS)
* 2-minute walk test

Data analysis:

As a pilot study, 20 children will be recruited for this study. Independent t-test or Mann Whitney U test will be used to compare the continuous and ordinal results between the intervention and control groups.

Expected results:

The trunk control, balance and gross motor function of children with CP will be significantly improved after the intervention.

Clinical significance and potential of the study:

This is clinical trial to examine the effectiveness of a new intervention, a kind of interactive computer play training module, on training the trunk control for children with cerebral palsy. If the intervention is proven effective, it may be an adjunct to the conventional Physiotherapy to children with movement disorders in enhancing their trunk control. Better trunk control will in turn improve the daily function for these children as their sitting and standing balance is improved. In a long run, these children will not rely on expensive seating equipment to maintain their balance during schooling and at home.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common physical disabilities in childhood, affecting 2 to 2.5 per 1000 live-births worldwide and about 1.3 per 1000 live-births in Hong Kong. It is a non-progressive lesion of the developing central nervous system affecting the control of movements and postures in the children. Children with CP are usually classified using the Gross Motor Function Classification System (GMFCS) according to age-specific gross motor functional abilities and reliance on assistive devices (such as walking aids or wheeled mobility). It is an ordinal grading system of five levels (I to V), in which self-initiated movements, such as sitting, standing or walking, are described in relation to different age groups. Children of levels I and II can generally walk without aids while children of level III can walk with aids for short distances but usually choose wheeled mobility in community settings. Children at level IV have limited motor ability in assisted standing, stepping, and transfers. Children classified as level V are completely dependent for transportation in a wheelchair and lack antigravity postural control. Numerous studies have shown that children with CP, regardless their GMFCS levels, demonstrate problems in their postural control in sitting and standing, which in turn affect their function and participation in daily life. The main deficits in postural control in sitting for children with CP are lack of ability to recruit direction-specific muscles in more severe children (GMFCS levels IV and V) or inability to fine-tune the degree of muscle contraction according to specific situations. Excessive contraction of antagonists is a common compensatory strategy. These ineffective strategies to compensate their balance in sitting or standing positions will affect the children's daily function such as desk work at school, transfers and ambulation.

Postural control involves controlling the body's position in space for stability and motility. Good postural control around the trunk or 'trunk control' in short, allows an individual to perform different tasks in an upright and vertical posture without losing the balance. The control of trunk to maintain balance in either sitting or standing positions is usually tested in the following three conditions: static balance, anticipatory balance and reactive balance. Assessment of trunk control in children is commonly part of a motor assessment such as Bruininks-Osteretsky Test of Motor Proficiency. The main limitation of these motor assessments is that the trunk is considered a one unit during a motor act, despite that there are different segments in the spine. Preliminary findings in very young infants have shown that infants with lumbar control had better movement quality in reaching actions when compared to those with thoracic control only. It seems that specific outcome measures on trunk control are necessary to demonstrate improvement in movement quality like this. There are specific outcome measures assessing balance, an indication of trunk control in recovering stability after internal or external perturbations such as Pediatric Reach Test (PRT), Pediatric Balance Scale, and Segmental Assessment on Trunk control (SATCo). It has been found very few of the commonly used outcome measures on balance have covered assessing all three aspects of balance as mentioned above. Most of these outcome measures require the children to be able to sit independently with or without hand support, making it unsuitable for children with CP of GMFCS levels IV and V. Furthermore, most of these outcome measures have the same limitation in considering the trunk as one whole unit, not consisting of different regions. Among all the commonly used assessment of trunk control, SATCo is a recently refined assessment on segmental trunk control in children. The child's trunk control is examined by progressively reducing the trunk support from the shoulder girdle to the pelvis in order to assess the head control, upper thoracic, mid-thoracic, lower thoracic, upper lumbar, lower lumbar and full trunk control. The trunk control is tested under 3 different conditions in sitting: to maintain the posture (static control), during voluntary head movements (active control) and recovery of trunk control after a disturbance of balance by a nudge (reactive control). (Butler et al, 2010) The preliminary results of the SATCo showed a high inter-rater reliability (ICC ≥ 0.8) and moderate to good correlations with other established motor assessments (r from 0.65 to 0.88). Besides assessing the trunk in different segments, SATCO is one of the rare ones being able to assess reactive balance. It has been recommended that to increase the comprehensiveness in assessing the balance mechanism in children with CP, researchers can use the SATCo in combination of outcome measures assessing more dynamic sitting balance, such as the PRT.

Interactive computer play (ICP) has become popular in rehabilitation for people with motor impairments, including children with CP. During an ICP, a child interacts and plays with virtual objects in a computer-generated environment, through the use of a computer console or platform and the software, allowing the child to control the games through certain body movements. Because the computer games are fun and enjoyable, the child will repeat the required body movements in numerous times so as to get a high score in the game without losing the interest. These numerous repetitions (essentially mass practice) and feedback from the game scores (knowledge of performance and results) are important in motor learning and enhancing neuroplasticity. Hence, ICP may be a feasible way to improve trunk control in children with CP, in addition to the conventional therapies. Up to date, there are six published studies using ICP or virtual reality in improving balance in children with CP.. From these 6 published studies, promising though conflicting results were found whether ICP is effective in improving trunk control in children with CP. The main limitations of these studies are the overall low levels of study quality, small sample sizes and heterogeneous population groups under the umbrella term CP. In fact, similar conclusions for future studies with larger sample sizes and rigorous study designs have been echoed from the four recent systematic reviews on the topic.

One of possible reasons for the conflicting conclusion on the use of ICP in rehabilitation for children with CP may be lack of sensitive outcome measures to capture the specific changes in the trunk control post-intervention. The above-mentioned studies were either using general motor assessments or outcome measures with unknown psychometric properties to assess the posture of the participants. Besides, when the child received the ICP intervention in a standing position, compensatory strategies, due to uncontrolled degrees of freedom in lower limbs, might be used to maintain their trunk control in this more challenging position than a sitting position. These compensatory strategies may in turn, water down the overall effect of the ICP intervention on the trunk control. Most of these studies examined only one or two aspect of the trunk control as testing the static or anticipatory balance of the children. The commercial gaming consoles, such as Nintendo Wii Fit, are not specifically developed for children with CP to elicit targeted movements to overcome their impairment and the software may not be sensitive enough to translate the subtle movement changes to an increase in the game scores as well to an adequate challenge for these children.

Tymo (Tyromotion, Austria, www.tyromotion.com) is a wireless force plate detecting the movement of the centre of pressure, either in a sitting or standing position. Force and weight distribution can be measured using the software provided with the Tymo in these two positions. During the assessment, the user will move the trunk forward, backward and sideways as far as they can. The amplitude of the force and weight distribution between the two sides of the body will be recorded. This information will be used when the user uses the Tymo as a balance training module, in which the user will move the trunk forward, backward and sideways to participate in a computer game. For example, the user will move their trunk in different directions so as to manoeuvre a basket to catch the falling apples. The difficulties of the game will be adjusted according to the information provided during the assessment so that the user needs to move their body accordingly in different directions without losing their balance. This equipment is specially designed for rehabilitation for people with movement disorders, hence unlike the commercial games, there are no flashing lights or sudden noises during the games.

20 children with CP or similar physical disabilities will be recruited from 2 special schools for children with physical disabilities in Hong Kong. Informed consent will be sought from the parents or guardians before the study will commence. After the initial assessment, all study children will be randomly allocated into a control group or treatment group (10 children in each arm) using a 'draw card from the hat'. The randomization will be separately done in each school. The children in the treatment group will receive training on their trunk control using the Tymo in sitting 4 times per week for 20 minutes per session. The treatment will last for 6 weeks. All study children will continue their usual therapies at school but will be asked to stop playing any interactive computer play, which is designed to train balance such as Nintendo Wii balance board, during the study period. As there is no strong research evidence that commercial computer games are effective in improving the balance for children with CP and this type of commercial computer play is not a routine training exercises for balance at the schools, it is believed that discontinuing this type of 'training' for 6 weeks would not cause detrimental effect on the balance of the study children.

All the assessment will be carried out by a blinded assessor, who is not aware of the group allocation of the children. All the children will be assessed at the beginning, and 3, 6 and 12 weeks after the commencement of the intervention.

All children will be calibrated using the Tymo in a static sitting position in each treatment session by the research staff and the amplitude of the force and weight distribution generated by the child between the two sides of the body will be recorded. This information will be used to set up the Tymo as a training module (the intervention) by the software, in which the child will move the trunk forward, backward and sideways to participate in a computer game in sitting. The child will choose which game they want in each treatment session and they have to stay on the same game for at least 10 minutes before changing to another game. The child will have a maximal choice of 2 computer games in each treatment session. All children will start at a medium level of difficulty. Only if the child is unable to score any point in 3 trials in a row, the difficulty level will be reduced to one level down. Similarly, if the child scores full points in 3 trials in a row, the difficulty level will be increased to one level up. The progression of the intervention will then be closely monitored by the research staff. A logbook will be used for each child to record the level of difficulty in each treatment session, the number of treatment sessions, duration of each session and general comments on the child in each session during the intervention phase by a research assistant.

ELIGIBILITY:
Inclusion Criteria:

1. Children with a diagnosis of CP will be of GMFCS levels III to IV, who in general, require walking aid (level III) during ambulation and with limited walking ability (level IV).[4] Aiming to achieve a higher homogeneity of the recruited children, for those with level III, only those requiring physical assistance to climb stairs will be recruited and so it is believed that only those with lower motor ability, i.e. similar to level IV, will be included.
2. Children, with non-CP physical disabilities, will have similar gross motor function as in (1).
3. Aged from 6 to 12 years old and
4. Able to follow instructions to interact in simple computer games

Exclusion Criteria:

Children with epilepsy/ seizures that could be elicited by flashing lights or sudden loud noises from computer screens

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamis W Pin, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oskoui M, Coutinho F, Dykeman J, Jette N, Pringsheim T. An update on the prevalence of cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2013 Jun;55(6):509-19. doi: 10.1111/dmcn.12080. Epub 2013 Jan 24. PMID 23346889
- [Background] Yam WK, Chan HS, Tsui KW, Yiu BP, Fong SS, Cheng CY, Chan CW; Working Group on Cerebral Palsy, Hong Kong Society of Child Neurology and Developmental Paediatrics. Prevalence study of cerebral palsy in Hong Kong children. Hong Kong Med J. 2006 Jun;12(3):180-4. PMID 16760544
- [Background] Mutch L, Alberman E, Hagberg B, Kodama K, Perat MV. Cerebral palsy epidemiology: where are we now and where are we going? Dev Med Child Neurol. 1992 Jun;34(6):547-51. doi: 10.1111/j.1469-8749.1992.tb11479.x. No abstract available. PMID 1612216
- [Background] Palisano R, Rosenbaum P, Walter S, Russell D, Wood E, Galuppi B. Development and reliability of a system to classify gross motor function in children with cerebral palsy. Dev Med Child Neurol. 1997 Apr;39(4):214-23. doi: 10.1111/j.1469-8749.1997.tb07414.x. PMID 9183258
- [Background] Butler PB, Saavedra S, Sofranac M, Jarvis SE, Woollacott MH. Refinement, reliability, and validity of the segmental assessment of trunk control. Pediatr Phys Ther. 2010 Fall;22(3):246-57. doi: 10.1097/PEP.0b013e3181e69490. PMID 20699770
- [Background] Rachwani J, Santamaria V, Saavedra SL, Wood S, Porter F, Woollacott MH. Segmental trunk control acquisition and reaching in typically developing infants. Exp Brain Res. 2013 Jul;228(1):131-9. doi: 10.1007/s00221-013-3544-y. Epub 2013 May 17. PMID 23681292
- [Background] Banas BB, Gorgon EJ. Clinimetric properties of sitting balance measures for children with cerebral palsy: a systematic review. Phys Occup Ther Pediatr. 2014 Aug;34(3):313-34. doi: 10.3109/01942638.2014.881952. Epub 2014 Feb 3. PMID 24490854
- [Background] Fehlings D, Switzer L, Findlay B, Knights S. Interactive computer play as "motor therapy" for individuals with cerebral palsy. Semin Pediatr Neurol. 2013 Jun;20(2):127-38. doi: 10.1016/j.spen.2013.06.003. PMID 23948687
- [Background] Sandlund M, McDonough S, Hager-Ross C. Interactive computer play in rehabilitation of children with sensorimotor disorders: a systematic review. Dev Med Child Neurol. 2009 Mar;51(3):173-9. doi: 10.1111/j.1469-8749.2008.03184.x. Epub 2009 Jan 26. PMID 19191834
- [Background] Snider L, Majnemer A, Darsaklis V. Virtual reality as a therapeutic modality for children with cerebral palsy. Dev Neurorehabil. 2010;13(2):120-8. doi: 10.3109/17518420903357753. PMID 20222773
- [Background] Deutsch JE, Borbely M, Filler J, Huhn K, Guarrera-Bowlby P. Use of a low-cost, commercially available gaming console (Wii) for rehabilitation of an adolescent with cerebral palsy. Phys Ther. 2008 Oct;88(10):1196-207. doi: 10.2522/ptj.20080062. Epub 2008 Aug 8. PMID 18689607
- [Background] Jelsma J, Pronk M, Ferguson G, Jelsma-Smit D. The effect of the Nintendo Wii Fit on balance control and gross motor function of children with spastic hemiplegic cerebral palsy. Dev Neurorehabil. 2013;16(1):27-37. doi: 10.3109/17518423.2012.711781. Epub 2012 Oct 3. PMID 23030836
- [Background] Ramstrand N, Lygnegard F. Can balance in children with cerebral palsy improve through use of an activity promoting computer game? Technol Health Care. 2012;20(6):501-10. doi: 10.3233/THC-2012-0696. PMID 23187015
- [Background] Sharan D, Ajeesh PS, Rameshkumar R, Mathankumar M, Paulina RJ, Manjula M. Virtual reality based therapy for post operative rehabilitation of children with cerebral palsy. Work. 2012;41 Suppl 1:3612-5. doi: 10.3233/WOR-2012-0667-3612. PMID 22317271
- [Background] Wade W, Porter D. Sitting playfully: does the use of a centre of gravity computer game controller influence the sitting ability of young people with cerebral palsy? Disabil Rehabil Assist Technol. 2012 Mar;7(2):122-9. doi: 10.3109/17483107.2011.589485. Epub 2011 Oct 4. PMID 21967300
- [Background] Bartlett D, Birmingham T. Validity and reliability of a pediatric reach test. Pediatr Phys Ther. 2003 Summer;15(2):84-92. doi: 10.1097/01.PEP.0000067885.63909.5C. PMID 17057438
- [Background] Pin TW. Psychometric properties of 2-minute walk test: a systematic review. Arch Phys Med Rehabil. 2014 Sep;95(9):1759-75. doi: 10.1016/j.apmr.2014.03.034. Epub 2014 May 9. PMID 24814460

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: The children in the treatment group will receive training on their trunk control using the Tymo in sitting 4 times per week for 20 minutes per session. The treatment will last for 6 weeks. All study children will continue their usual therapies at school.
  Tymo: All children will be calibrated using the Tymo in a static sitting position in each treatment session. The amplitude of the force and weight distribution generated by the child between the two sides of the body will be recorded. This information will be used to set up the Tymo as a training module (the intervention) by the software, in which the child will move the trunk forward, backward and sideways to participate in a computer game in sitting. The child will choose which game they want in each treatment session and they have to stay on the same game for at least 10 minutes before changing to another game.
- Control: Children in the control group will continue their usual therapy.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: the analysis population was not different from the assignment in the Participant Flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 18
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.92 (2.25) | 9.59 (1.87) | 9.26 (2.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 5 | 6 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Segmental Assessment on Trunk Control-static
Description: assess the level of static segmental trunk control. Assessment score represents as follows: 1= learning head control, 2= learning upper thoracic control, 3= learning mid-thoracic control, 4= learning lower thoracic control, 5= learning at upper lumber control, 6= learning lower lumbar control, 7= learning full trunk control and 8= achieved full trunk control.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 8 [7 to 8] | 8 [5 to 8]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Segmental Assessment on Trunk Control-active
Description: assess the level of active segmental trunk control. Assessment score represents as follows: 1= learning head control, 2= learning upper thoracic control, 3= learning mid-thoracic control, 4= learning lower thoracic control, 5= learning at upper lumber control, 6= learning lower lumbar control, 7= learning full trunk control and 8= achieved full trunk control.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 7 [5 to 8] | 8 [4 to 8]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Segmental Assessment on Trunk Control-reactive
Description: assess the level of reactive segmental trunk control. Assessment score represents as follows: 1= learning head control, 2= learning upper thoracic control, 3= learning mid-thoracic control, 4= learning lower thoracic control, 5= learning at upper lumber control, 6= learning lower lumbar control, 7= learning full trunk control and 8= achieved full trunk control.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 6 [4 to 8] | 6 [1 to 8]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Pediatric Reach Test-forward Sitting
Description: assess how far the child can reach forward in sitting
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Intervention | Control
Number analyzed (Participants) | 9 | 9
centimeters | 8.28 (74.5) | 10.72 (96.5)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, t-test, 2 sided

5. Secondary Outcome: Pediatric Reach Test- Right Sitting
Description: assess how far the child can reach to his/her right in sitting
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Intervention | Control
Number analyzed (Participants) | 9 | 9
centimeters | 8.5 (76.5) | 10.5 (94.5)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, t-test, 2 sided

6. Secondary Outcome: Pediatric Reach Test- Left Sitting
Description: assess how far the child can reach to his/her left in sitting
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Intervention | Control
Number analyzed (Participants) | 9 | 9
centimeters | 8.94 (80.50) | 10.06 (90.50)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, t-test, 2 sided

7. Secondary Outcome: Pediatric Reach Test- Forward Standing
Description: assess how far the child can reach forward in standing
Time Frame: 12 weeks
Population: This outcome measure was abandoned as all the participants were unable to stand unaided long enough to complete the measurement.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Pediatric Reach Test- Right Standing
Description: assess how far the child can reach to his/her right in standing
Time Frame: 12 weeks
Population: as for outcome 7
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Pediatric Reach Test- Left Standing
Description: assess how far the child can reach to his/her left in standing
Time Frame: 12 weeks
Population: as for outcome 7
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Gross Motor Function Measure Item Set- Total Score
Description: assess the gross motor function using Gross Motor Function Measure Item Set.There are 4 Item Sets: Item Set 1 includes 15 test items (score ranged from 0 to 45), Item Set 2 including 29 items (score ranged from 0 to 87), Item Set 3 including 39 items (score ranged from 0 to 117) and Item Set 4 including 22 test items (score ranged from 0 to 66). Each participant will only be assessed with 1 Item Set based on their score on pre-defined decision items (Russell et al.Gross Motor Function Measure (GMFM-66 & GMFM-88) User's manual 2nd Edition. 2013). Individual item scores of the Item Set are entered and a mathematical algorithm calculates an interval level total score ranged from 0 to 100) using the Gross Motor Ability Estimator (GMAE-2) Scoring Software (https://www.canchild.ca/en/resources/191-gross-motor-ability-estimator-gmae-2-scoring-software-for-the-gmfm). The higher scores mean higher abilities.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 9 | 9
score on a scale | 9.06 (81.5) | 9.94 (89.5)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, t-test, 2 sided

11. Secondary Outcome: 2-minute Walk Test
Description: measure how far the study participant can walk in 2 minutes in metres
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Intervention | Control
Number analyzed (Participants) | 9 | 9
meters | 8.11 (73.0) | 10.89 (98.0)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, t-test, 2 sided

12. Secondary Outcome: Height
Description: measure the height of study participants in centimetres
Time Frame: 12 weeks
Population: Data was not collected in the study as it was determined that measurement of height was not related to any of the primary outcomes. To cut down this outcome measure could also reduce the unnecessary measurement burden on the study participants.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Weight
Description: measure the body weight of study participants in kilograms
Time Frame: 12 weeks
Population: Data was not collected in the study as it was determined that measurement of weight was not related to any of the primary outcomes. To cut down this outcome measure could also reduce the unnecessary measurement burden on the study participants.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Gross Motor Function Measure 88- Lying
Description: assess the gross motor function in lying and rolling using Gross Motor Function Measure 88-lying (score ranged from 0 to 51) where higher score means higher gross motor function in this position.
Time Frame: 12 weeks
Population: This outcome has been abandoned as it was decided to use a concise version of Gross Motor Function Measure Item Set to avoid over-burdening of the study participants.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Gross Motor Function Measure 88- Sitting
Description: assess the gross motor function inlsitting using Gross Motor Function Measure 88-sitting (score ranged from 0 to 60) where higher score means higher gross motor function in this position.
Time Frame: 12 weeks
Population: as for outcome 14
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Gross Motor Function Measure 88- Crawling and Kneeling
Description: assess the gross motor function in crawling position using Gross Motor Function Measure 88-crawling and kneeling (score ranged from 0 to 42) where higher score means higher gross motor function in this position.
Time Frame: 12 weeks
Population: as for outcome 14
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Gross Motor Function Measure 88- Standing
Description: assess the gross motor function in standing position using Gross Motor Function Measure 88-standing (score ranged from 0 to 39) where higher score means higher gross motor function in this position.
Time Frame: 12 weeks
Population: as for outcome 14
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
1. Children should have a reasonable level of cognitive function to participate in the interactive computer play. Cognitive impairment is a common co-morbidities.
2. Small sample size
3. Increase type 1 error as repeated measurements on participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT02975804/Prot_SAP_000.pdf